CLINICAL TRIAL: NCT04796038
Title: Evaluation of the Acute Safety and Device Success of the RISE SC Coronary Balloon Dilatation Catheter When Used as a Dilatation Device in the Stenotic Portion of a Coronary Artery or Bypass Graft in Patients With Coronary Artery Disease
Brief Title: Rise Semi Compliant Balloon Study in Patient With CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-EU-02
Record Dates: First submitted 2021-02-10; First posted 2021-03-12 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rise SC (Experimental): All patients will receive the Rise semi-compliant balloon catheter as per treatment.
  Interventions: Device: Balloon dilatation

INTERVENTIONS:
Device: Balloon dilatation — Patient will be treated with balloon dilatation either stand-alone (POBA) or followed by stent implantation.

SUMMARY:
Single arm, prospective, multi-center, trial designed to enrol approximately 66 patients. All patients will undergo PCI using at least one RISE SC balloon as per routine clinical practice and will be followed until discharge for data collection. Patients will be enrolled in up to 5 investigational sites in Switzerland.

The patients will be followed up until discharge or until 7 days, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria

  1. Subject must be at least 18 years of age.
  2. Subject or a legally authorised representative must provide written informed consent prior to any study related procedure.
  3. Subject must have stenotic lesion(s) in native coronary arteries or bypass grafts that are suitable for percutaneous coronary intervention.
  4. Subject must agree to undergo all protocol-required follow-up procedures.
  5. Subject must agree not to participate in any other clinical study during hospitalisation for the index procedure.
* Angiographic Inclusion Criteria All angiographic inclusion criteria are based on visual estimation.

  1. De novo or restenotic lesions in native coronary arteries or bypass grafts.
  2. A maximum of two lesions, with either both in one vessel or one lesion in each of two vessels.
  3. The target lesion(s) must have a diameter stenosis of ≥ 50% by visual estimation or online quantitative coronary angiography (QCA) and may include chronic total occlusions (CTO).

Exclusion Criteria:

* General Exclusion Criteria

  1. Planned use of a non-study angioplasty balloon during the procedure for pre-dilatation or dilatation of the lesion.
  2. Subject has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, other anti-platelet medications, or sensitivity to contrast media, which cannot be adequately pre-treated.
  3. Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3.
  4. Subject is currently participating in an investigational study that may confound the treatment or outcomes of this study.
  5. Subject is pregnant or nursing. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.
* Angiographic Exclusion Criteria All angiographic exclusion criteria are based on visual estimation.

  1. Unprotected left main coronary artery disease
  2. More than two lesions requiring treatment. Tandem lesions, defined as multiple, focal lesions that can be covered by one balloon, will be considered as a single lesion.
  3. Coronary artery spasm in the absence of significant stenosis.
  4. Anticipated need for plaque modification using rotational/orbital atherectomy or intravascular lithotripsy. Note: The use of scoring or cutting balloons after (pre)-dilatation with the study device is allowed.
  5. Additional clinically significant lesion(s) in any coronary arteries or bypass grafts for which PCI may be required during hospitalization for the index procedure (in-hospital staged PCI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Percentage of treated lesions with device success defined as: | During the interventional procedure
  1. Successful device delivery and
  2. Successful inflation and deflation of the balloon and
  3. No perforation, flow-limiting dissection or reduction in TIMI flow grade and
  4. No life-threatening arrhythmias (sustained Ventricular Tachycardia (VT), Ventricular Fibrillation (VF))

SECONDARY OUTCOMES:
Percentage of patients with Individual components of device success defined as: | During the interventional procedure
  1. Successful device delivery
  2. Successful inflation and deflation of the balloon
  3. No perforation, flow-limiting dissection or reduction in TIMI flow grade
  4. No life-threatening arrhythmias (sustained VT, VF)
Percentage of patients with Procedural success defined as: | 1 - 7 Days
  Device success without major adverse cardiovascular events (MACE) which is a composite of all death, myocardial infarction (MI), and clinically indicated target lesion revascularization (CI-TLR) by coronary artery bypass graft surgery (CABG) or percutaneous coronary intervention (PCI) during the index hospitalization.
Percentage of patients with Target Lesion Failure (TLF) | 1 - 7 Days
  A composite of cardiac death, target vessel myocardial infarction (TV-MI), and CI-TLR by CABG or PCI during the index hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Roffi, Dr., Principal Investigator — Hôpitaux universitaires de Genève (HUG)
Locations (3):
- Switzerland (3):
  - CHUV, Lausanne, Canton of Vaud
  - HVS, Sion, Valis
  - HUG, Geneva

IPD SHARING:
Plan to Share IPD: Yes
The emphasis in all scientific publications and presentations will be placed on the endpoint at discharge.